CLINICAL TRIAL: NCT07266922
Title: Running Informed, Not Just Trained: A Self-Directed Web-Based Education for Boston Marathon Runners With Patellofemoral Pain
Brief Title: A Self-Directed Web-Based Education for Boston Marathon Runners With Patellofemoral Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sungwan Kim, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00052732
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Patellofemoral Pain
Keywords: Anterior knee pain; Patient education
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: We will conduct a two-arm, parallel-group, single-blinded randomized controlled trial to evaluate the effect of the intervention prior to the marathon (Group 1: treatment vs. Group 2: wait-and-see control). After the marathon, Group 2 will receive the same intervention, and outcomes will be assessed in a quasi-experimental pre-post design (i.e., as a single treatment group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Marathon Education (Experimental): This group will receive the educational platform for 6 weeks prior to the 2026 Boston Marathon. Participants will have access to MyKneeCap.com, a web-based platform designed to provide runners with evidence-based education on the physical and non-physical factors contributing to patellofemoral pain, as well as strategies for self-managing symptoms tailored specifically for runners.
  Interventions: Behavioral: Education Platform-MyKneeCap.com
- Wait-and-See Control / Post-Marathon Education (Other): This group will serve as a wait-and-see control (no intervention) prior to the 2026 Boston Marathon. After completing the marathon, participants will receive access to MyKneeCap.com, a web-based platform designed to provide runners with evidence-based education on the physical and non-physical factors contributing to patellofemoral pain, as well as strategies for self-managing symptoms tailored specifically for runners.
  Interventions: Behavioral: Education Platform-MyKneeCap.com

INTERVENTIONS:
Behavioral: Education Platform-MyKneeCap.com — This intervention uses MyKneeCap.com, a free, web-based educational platform designed to help runners understand their knee pain. The platform provides information about patellofemoral pain and includes exercise programs aimed at reducing pain and improving knee function. This intervention does not involve any drugs, devices, or other procedural components.

SUMMARY:
Runners experience diverse lower extremity injuries, and the most common is patellofemoral pain (PFP)-commonly known as "runner's knee" and characterized by pain around and/or behind the kneecap. The aim of this study is to evaluate the effectiveness of a 6-week, self-directed, web-based education program for runners competing in the 2026 Boston Marathon. The study will evaluate outcomes, including pain, function, and marathon performance, in runners who use a web-based educational program designed to help them understand and manage knee pain. There will be two groups: Group 1 will receive the 6-week web-based educational program prior to the 2026 Boston Marathon, while Group 2 will serve as the wait-and-see control group (no intervention) prior to the marathon and then receive the same program 6 weeks after completing the marathon.

ELIGIBILITY:
Inclusion Criteria:

* Insidious onset of peripatellar and/or retropatellar pain ≥3 months
* Worst pain level in the previous week ≥3/10 on the numeric pain rating scale
* Pain during at least two of the following tasks: prolonged sitting, kneeling, squatting, walking, running, jumping, and stair negotiation.
* All participants must have access to an internet-enabled device (e.g., computer, tablet, smartphone) equipped with audio capabilities sufficient to engage with the web-based education platform

Exclusion Criteria:

* History of lower extremity surgery
* History of lower extremity pain or injury (other than patellofemoral pain) in the previous six months
* History of patellar dislocation or subluxation
* Internal derangement (e.g., meniscal lesion)
* Ligamentous instability
* Other sources of anterior knee pain (e.g., patellar tendinopathy, bursitis)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes (pain) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Pain will be assessed for current pain and worst pain in the previous week using a 10-cm visual analog scale (VAS; 0=no pain; 10=worst pain imaginable), a reliable, valid, and responsive tool for evaluating treatment outcomes for patellofemoral pain.
Clinical outcomes (self-reported function) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Self-reported function will be evaluated using the 11-item Knee Injury and Osteoarthritis Outcome Score-Patellofemoral subscale (KOOS-PF; 0=extreme disability; 100=no disability), a reliable tool with the highest content validity for patellofemoral pain.
Clinical outcomes (global rating of change) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Global rating of change will be assessed for perceived recovery using a 7-point Likert scale (much worse, worse, slightly worse, no change, slightly better, better, or much better). The global rating of change scale is a reliable, clinically relevant, and patient-centered measure for interpreting meaningful improvements.

SECONDARY OUTCOMES:
Psychological function (fear-avoidance beliefs) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Fear-avoidance beliefs will be quantified using the 5-item Fear-Avoidance Beliefs Questionnaire-Physical Activity subscale (FABQ-PA; 0=no fear-avoidance; 24=extreme fear-avoidance). The FABQ-PA is a reliable and valid tool and represents a key psychological profile in patellofemoral pain management.
Psychological function (pain self-efficacy) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Pain self-efficacy will be quantified using the 10-item Pain Self-Efficacy Questionnaire (PSEQ; 0=no self-efficacy; 60=extreme self-efficacy). The PSEQ is a reliable and valid tool and represents a key psychological profile in patellofemoral pain management.
Patient satisfaction | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Satisfaction during the preceding six weeks of marathon training will be rated on a 5-point Likert scale (very dissatisfied, somewhat dissatisfied, neither, somewhat satisfied, or very satisfied).
Marathon performance (finish time) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Finish time will be evaluated by comparing the official finish time to the participant's intended finish time (in minutes).
Marathon performance (division ranking) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Division ranking will be evaluated by comparing the division ranking to the participant's intended division ranking (in rank).
Medical service use | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Intra-event medical encounters for knee pain will be self-recorded (in count).
Secondary musculoskeletal complaints | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Lower extremity pain or injuries (other than patellofemoral pain) sustained during the race will be self-recorded (in count).
Return to running readiness | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Perceived readiness to return to competitive running will be assessed on a 5-point Likert scale (not at all, slightly, moderately, very, or extremely).
Barriers and facilitators (confidence in self-management) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Confidence in self-management ("I am confident in my ability to manage my symptoms and treatment plan on my own") will be measured using a 5-point Likert scale (strongly disagree, disagree, neither, agree, strongly agree).
Barriers and facilitators (usability of the education platform) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Usability of the education platform ("The web-based education platform is easy to use and navigate") will be measured using a 5-point Likert scale (strongly disagree, disagree, neither, agree, strongly agree).
Barriers and facilitators (treatment expectations) | 6-weeks leading up to the Boston Marathon, or 6-weeks post completion of Boston Marathon
  Treatment expectations ("I believe that the web-based education and exercise program will help improve my condition") will be measured using a 5-point Likert scale (strongly disagree, disagree, neither, agree, strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Sungwan Kim, PhD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
All IPD that will be shared will be de-identified and for manuscript and publishing purposes only. PHI data will not be accessible outside of the research team, and only de-identified data will be a part of the manuscript.
Time Frame: IPD will be analyzed for the manuscript, and all will be de-identified. This is approximately from the end of the study collection June 2026 to September 2026 for analysis.

REFERENCES:
- [Background] Piva SR, Gil AB, Moore CG, Fitzgerald GK. Responsiveness of the activities of daily living scale of the knee outcome survey and numeric pain rating scale in patients with patellofemoral pain. J Rehabil Med. 2009 Feb;41(3):129-35. doi: 10.2340/16501977-0295. PMID 19229444
- [Background] Evans JD. Straightforward statistics for the behavioral sciences. Thomson Brooks/Cole Publishing Co; 1996
- [Background] Cohen J. Statistical power analysis for the behavioral sciences. Academic press; 1988
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] Briggs KK, Lysholm J, Tegner Y, Rodkey WG, Kocher MS, Steadman JR. The reliability, validity, and responsiveness of the Lysholm score and Tegner activity scale for anterior cruciate ligament injuries of the knee: 25 years later. Am J Sports Med. 2009 May;37(5):890-7. doi: 10.1177/0363546508330143. Epub 2009 Mar 4. PMID 19261899
- [Background] Vicenzino BT, Rathleff MS, Holden S, Maclachlan L, Smith BE, de Oliveira Silva D, van Middelkoop M. Developing Clinical and Research Priorities for Pain and Psychological Features in People With Patellofemoral Pain: An International Consensus Process With Health Care Professionals. J Orthop Sports Phys Ther. 2022 Jan;52(1):29-39. doi: 10.2519/jospt.2022.10647. PMID 34972490
- [Background] Asghari A, Nicholas MK. Pain self-efficacy beliefs and pain behaviour. A prospective study. Pain. 2001 Oct;94(1):85-100. doi: 10.1016/S0304-3959(01)00344-X. PMID 11576748
- [Background] Piva SR, Fitzgerald GK, Irrgang JJ, Fritz JM, Wisniewski S, McGinty GT, Childs JD, Domenech MA, Jones S, Delitto A. Associates of physical function and pain in patients with patellofemoral pain syndrome. Arch Phys Med Rehabil. 2009 Feb;90(2):285-95. doi: 10.1016/j.apmr.2008.08.214. PMID 19236982
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Crossley KM, Macri EM, Cowan SM, Collins NJ, Roos EM. The patellofemoral pain and osteoarthritis subscale of the KOOS (KOOS-PF): development and validation using the COSMIN checklist. Br J Sports Med. 2018 Sep;52(17):1130-1136. doi: 10.1136/bjsports-2016-096776. Epub 2017 Mar 3. PMID 28258176
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407
- [Background] Souto LR, Pazzinatto MF, De Oliveira Silva D, Ezzat AM, Barton CJ. Self-directed versus supervised exercise therapy program combined with digitally supported patient education for knee osteoarthritis: a randomised, parallel-group feasibility trial. Semin Arthritis Rheum. 2025 Oct;74:152787. doi: 10.1016/j.semarthrit.2025.152787. Epub 2025 Jul 20. PMID 40716116
- [Background] Barton CJ, de Oliveira Silva D, Patterson BE, Crossley KM, Pizzari T, Nunes GS. A proximal progressive resistance training program targeting strength and power is feasible in people with patellofemoral pain. Phys Ther Sport. 2019 Jul;38:59-65. doi: 10.1016/j.ptsp.2019.04.010. Epub 2019 May 2. PMID 31055059
- [Background] Lack S, Neal B, De Oliveira Silva D, Barton C. How to manage patellofemoral pain - Understanding the multifactorial nature and treatment options. Phys Ther Sport. 2018 Jul;32:155-166. doi: 10.1016/j.ptsp.2018.04.010. Epub 2018 Apr 12. PMID 29793124
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] Barton CJ, Lack S, Hemmings S, Tufail S, Morrissey D. The 'Best Practice Guide to Conservative Management of Patellofemoral Pain': incorporating level 1 evidence with expert clinical reasoning. Br J Sports Med. 2015 Jul;49(14):923-34. doi: 10.1136/bjsports-2014-093637. Epub 2015 Feb 25. PMID 25716151
- [Background] Liao TC, Keyak JH, Powers CM. Runners With Patellofemoral Pain Exhibit Greater Peak Patella Cartilage Stress Compared With Pain-Free Runners. J Appl Biomech. 2018 Aug 1;34(4):298-305. doi: 10.1123/jab.2017-0229. Epub 2018 Jul 11. PMID 29485362
- [Background] Bazett-Jones DM, Cobb SC, Huddleston WE, O'Connor KM, Armstrong BS, Earl-Boehm JE. Effect of patellofemoral pain on strength and mechanics after an exhaustive run. Med Sci Sports Exerc. 2013 Jul;45(7):1331-9. doi: 10.1249/MSS.0b013e3182880019. PMID 23377834
- [Background] Willy RW, Hoglund LT, Barton CJ, Bolgla LA, Scalzitti DA, Logerstedt DS, Lynch AD, Snyder-Mackler L, McDonough CM. Patellofemoral Pain. J Orthop Sports Phys Ther. 2019 Sep;49(9):CPG1-CPG95. doi: 10.2519/jospt.2019.0302. PMID 31475628
- [Background] Silva DDO, Pazzinatto M, Azevedo F, Crossley K, Barton C. Web-based multimedia education for people with patellofemoral pain: a preliminary analysis of a randomised controlled trial. J Sci Med Sport. 2018;21:S52-S53.
- [Background] De Oliveira Silva D, Pazzinatto MF, Crossley KM, Azevedo FM, Barton CJ. Novel Stepped Care Approach to Provide Education and Exercise Therapy for Patellofemoral Pain: Feasibility Study. J Med Internet Res. 2020 Jul 22;22(7):e18584. doi: 10.2196/18584. PMID 32706674
- [Background] Esculier JF, Maggs K, Maggs E, Dubois B. A Contemporary Approach to Patellofemoral Pain in Runners. J Athl Train. 2020 Nov 16;55(12):0. doi: 10.4085/1062-6050-0535.19. PMID 33196837
- [Background] Smith BE, Moffatt F, Hendrick P, Bateman M, Rathleff MS, Selfe J, Smith TO, Logan P. The experience of living with patellofemoral pain-loss, confusion and fear-avoidance: a UK qualitative study. BMJ Open. 2018 Jan 23;8(1):e018624. doi: 10.1136/bmjopen-2017-018624. PMID 29362256
- [Background] Maclachlan LR, Collins NJ, Matthews MLG, Hodges PW, Vicenzino B. The psychological features of patellofemoral pain: a systematic review. Br J Sports Med. 2017 May;51(9):732-742. doi: 10.1136/bjsports-2016-096705. Epub 2017 Mar 20. PMID 28320733
- [Background] Feely C, Smyth B, Caulfield B, Lawlor A. Estimating the cost of training disruptions on marathon performance. Front Sports Act Living. 2023 Jan 10;4:1096124. doi: 10.3389/fspor.2022.1096124. eCollection 2022. PMID 36704260
- [Background] Kim S, Wu Y, Glaviano NR, Pescatello LS. Physical Activity Levels in Persons With Patellofemoral Pain: A Systematic Review and Meta-analysis. Sports Health. 2025 Jul;17(4):804-814. doi: 10.1177/19417381241264494. Epub 2024 Aug 11. PMID 39129377
- [Background] Glaviano NR, Holden S, Bazett-Jones DM, Singe SM, Rathleff MS. Living well (or not) with patellofemoral pain: A qualitative study. Phys Ther Sport. 2022 Jul;56:1-7. doi: 10.1016/j.ptsp.2022.05.011. Epub 2022 May 26. PMID 35691244
- [Background] Blond L, Hansen L. Patellofemoral pain syndrome in athletes: a 5.7-year retrospective follow-up study of 250 athletes. Acta Orthop Belg. 1998 Dec;64(4):393-400. PMID 9922542
- [Background] Rathleff MS, Rathleff CR, Olesen JL, Rasmussen S, Roos EM. Is Knee Pain During Adolescence a Self-limiting Condition? Prognosis of Patellofemoral Pain and Other Types of Knee Pain. Am J Sports Med. 2016 May;44(5):1165-71. doi: 10.1177/0363546515622456. Epub 2016 Jan 20. PMID 26792702
- [Background] Glaviano NR, Baellow A, Saliba S. Physical activity levels in individuals with and without patellofemoral pain. Phys Ther Sport. 2017 Sep;27:12-16. doi: 10.1016/j.ptsp.2017.07.002. Epub 2017 Jul 18. PMID 28780340
- [Background] Holland AE. Telephysiotherapy: time to get online. J Physiother. 2017 Oct;63(4):193-195. doi: 10.1016/j.jphys.2017.08.001. Epub 2017 Sep 20. No abstract available. PMID 28939309
- [Background] Neal BS, Lack SD, Bartholomew C, Morrissey D. Best practice guide for patellofemoral pain based on synthesis of a systematic review, the patient voice and expert clinical reasoning. Br J Sports Med. 2024 Dec 18;58(24):1486-1495. doi: 10.1136/bjsports-2024-108110. PMID 39401870
- [Background] Souto LR, De Oliveira Silva D, Pazzinatto MF, Barton CJ. Beliefs of People With Patellofemoral Pain About Their Condition and Treatments Before and After Self-Directed Access to a Web-Based Education Platform. Musculoskeletal Care. 2025 Sep;23(3):e70165. doi: 10.1002/msc.70165. PMID 40736481
- [Background] de Oliveira Silva D, Pazzinatto MF, Rathleff MS, Holden S, Bell E, Azevedo F, Barton C. Patient Education for Patellofemoral Pain: A Systematic Review. J Orthop Sports Phys Ther. 2020 Jul;50(7):388-396. doi: 10.2519/jospt.2020.9400. Epub 2020 Apr 29. PMID 32349640
- [Background] Rathleff MS, Thomsen JL, Barton CJ. Patient education in patellofemoral pain: potentially potent and essential, but under-researched. Br J Sports Med. 2018 May;52(10):623-624. doi: 10.1136/bjsports-2017-098298. Epub 2017 Sep 19. No abstract available. PMID 28928114
- [Background] Crossley KM, van Middelkoop M, Callaghan MJ, Collins NJ, Rathleff MS, Barton CJ. 2016 Patellofemoral pain consensus statement from the 4th International Patellofemoral Pain Research Retreat, Manchester. Part 2: recommended physical interventions (exercise, taping, bracing, foot orthoses and combined interventions). Br J Sports Med. 2016 Jul;50(14):844-52. doi: 10.1136/bjsports-2016-096268. Epub 2016 May 31. No abstract available. PMID 27247098
- [Background] Taunton JE, Ryan MB, Clement DB, McKenzie DC, Lloyd-Smith DR, Zumbo BD. A retrospective case-control analysis of 2002 running injuries. Br J Sports Med. 2002 Apr;36(2):95-101. doi: 10.1136/bjsm.36.2.95. PMID 11916889
- [Background] Macintyre J, Taunton J, Clement D, Lloyd-Smith D, McKenzie D, Morrell R. Running injuries: a clinical study of 4,173 cases. Clin J Sport Med. 1991;1(2):81-87.
- [Background] Francis P, Whatman C, Sheerin K, Hume P, Johnson MI. The Proportion of Lower Limb Running Injuries by Gender, Anatomical Location and Specific Pathology: A Systematic Review. J Sports Sci Med. 2019 Feb 11;18(1):21-31. eCollection 2019 Mar. PMID 30787648
- [Background] Crossley KM, Stefanik JJ, Selfe J, Collins NJ, Davis IS, Powers CM, McConnell J, Vicenzino B, Bazett-Jones DM, Esculier JF, Morrissey D, Callaghan MJ. 2016 Patellofemoral pain consensus statement from the 4th International Patellofemoral Pain Research Retreat, Manchester. Part 1: Terminology, definitions, clinical examination, natural history, patellofemoral osteoarthritis and patient-reported outcome measures. Br J Sports Med. 2016 Jul;50(14):839-43. doi: 10.1136/bjsports-2016-096384. Epub 2016 Jun 24. No abstract available. PMID 27343241
- [Background] van Gent RN, Siem D, van Middelkoop M, van Os AG, Bierma-Zeinstra SM, Koes BW. Incidence and determinants of lower extremity running injuries in long distance runners: a systematic review. Br J Sports Med. 2007 Aug;41(8):469-80; discussion 480. doi: 10.1136/bjsm.2006.033548. Epub 2007 May 1. PMID 17473005
- [Background] van Mechelen W. Running injuries. A review of the epidemiological literature. Sports Med. 1992 Nov;14(5):320-35. doi: 10.2165/00007256-199214050-00004. PMID 1439399
- [Background] Hespanhol Junior LC, Pillay JD, van Mechelen W, Verhagen E. Meta-Analyses of the Effects of Habitual Running on Indices of Health in Physically Inactive Adults. Sports Med. 2015 Oct;45(10):1455-68. doi: 10.1007/s40279-015-0359-y. PMID 26178328
- [Background] Lee DC, Brellenthin AG, Thompson PD, Sui X, Lee IM, Lavie CJ. Running as a Key Lifestyle Medicine for Longevity. Prog Cardiovasc Dis. 2017 Jun-Jul;60(1):45-55. doi: 10.1016/j.pcad.2017.03.005. Epub 2017 Mar 30. PMID 28365296